CLINICAL TRIAL: NCT04932538
Title: Kinesio Taping On Gluteal Muscles: Does It Affect Balance, Functionality, And Participation In Children With Unilateral Spastic Cerebral Palsy?
Brief Title: Effects Of Kinesio Taping On Balance, Functionality, And Participation In Children With Cerebral Palsy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Seda Nur Kemer, Physiotherapist, Master of Science, Lecturer, Principal İnvestigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A7698
Record Dates: First submitted 2021-06-01; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Cerebral Palsy, Spastic; Gait Disorders, Neurologic; Hemiplegic Cerebral Palsy
Keywords: cerebral palsy; gait; balance; kinesio taping
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Every group received routine traditional physiotherapy twice a week over the period of 4 weeks. This routine traditional treatment consisted of stretching, weight bearing, functional reaching, walking, and electrotherapy.
- Kinesio Taping (Experimental): Every group received routine traditional physiotherapy twice a week over the period of 4 weeks. This routine traditional treatment consisted of stretching, weight bearing, functional reaching, walking, and electrotherapy. Sessions were 40 minutes. The children in the taping group were taped 6 days per week for 4 weeks. The children were checked for allergies before applying the tape. A 5-cm tape was applied and kept in position for 3 days, and the region was then left to rest for 24 hours.
  Interventions: Other: Kİnesio Taping

INTERVENTIONS:
Other: Kİnesio Taping — Kinesio Taping® (KT) is used for pediatric rehabilitation to reduce pain, facilitate or inhibit muscle activity, prevent injuries, reposition joints, aid the lymphatic system, support postural alignment, and improve proprioception
  Arms: Kinesio Taping

SUMMARY:
BACKGROUND: Walking and balance problems are among the most common problems in individuals with cerebral palsy (CP). Hip abduction and extension muscle function insufficiencies are common in children with CP.

OBJECTIVE: The aim of this study was to investigate the immediate and long-term effects of Kinesio® Taping (KT) applied on the gluteus maximus and gluteus medius muscles on walking, functionality, balance, and participation in children with unilateral spastic CP.

METHOD: This study was designed as a randomized controlled trial. The study included 20 children with unilateral spastic CP: 11 in the taping group and 9 in the control group. KT was applied in the taping group for 4 weeks in addition to a physiotherapy program. The control group received only the physiotherapy program. Body structure and functions were evaluated with the Pediatric Berg Balance Scale (PBBS). Activity was evaluated with the Timed Up and Go Test (TUG), Functional Mobility Scale (FMS), Gross Motor Function Scale (GMFM-88), the BTS G-Walk Spatiotemporal Gait Analysis System. Participation was evaluated with the Canadian Occupational Performance Measure (COPM). Evaluations were made at the beginning of the study and 30 minutes after the first tape application, and at the end of 4 weeks in the taping group. The level of significance was accepted as p<0.05.

DETAILED DESCRIPTION:
INTRODUCTION Walking and balance problems are frequently seen in individuals with cerebral palsy (CP). In individuals with CP, co-contraction of the distal and proximal muscles increase and muscle activation patterns are not fluent. Spasticity causes a decrease in muscle strength and length and a reduction in muscular coordination. Secondary to all this, decreases are seen in the energy production of the muscles.

Insufficiencies in hip abduction and extension muscle function are common in CP. Excessive muscles tonus in the hip adductors and flexors and a loss of reciprocal inhibition cause a weakness in the gluteus medius and maximus. This weakness negatively affects the movement patterns of the lumbar spine, pelvis, and hip region, and also causes incorrect loadings in hip joint and abnormalities in hip biomechanics. Gait anomalies occur and pelvis stabilization is impaired. In particular, negative impacts on participation are a concern. With the physiotherapy and rehabilitation approaches, these negative effects may be minimized by facilitating the gluteal muscles. Gait training and exercises to strengthen the gluteal muscles are routinely used in the rehabilitation of CP. With these approaches, it is aimed to maximize the gait function and promote independence and participation.

The somatosensory system may be affected in unilateral spastic CP. These children often suffer sensory impairments that could affect the development of future motor skills. Kinesio Taping® (KT) is used for pediatric rehabilitation to reduce pain, facilitate or inhibit muscle activity, prevent injuries, reposition joints, aid the lymphatic system, support postural alignment, and improve proprioception.

Yasukawa et al. stated that the use of KT for children with CP might influence the cutaneous receptors of the sensory motor system, resulting in an improvement in voluntary control and coordination via a physiotherapy program. Therefore, facilitating the gluteal muscles by KT may affect walking and balance positively.

In the literature, the clinical use of KT techniques in children with CP is generally at the upper extremity. In studies in which KT is applied to the lower extremity, it is generally applied to the distal part of extremity. In addition, most of the studies have investigated the immediate effect. There are few studies investigating the effects of KT applied to the gluteus medius and gluteus maximus muscles, which are located in the proximal hip with important contributions in stabilization.

The aim of this study was to investigate the immediate and long-term effects of KT applied to the gluteus maximus and gluteus medius muscles on walking, functionality, balance, and participation in children with unilateral spastic CP.

MATERIAL AND METHODS The permission of the University Ethics Committee was received (91610558-302.08.01) and written informed consent was obtained from each participant and/or guardian.

Participants

The inclusion criteria were: having unilateral spastic CP; being in an age between 6 years and 12 years; being classified in levels I or II of the Gross Motor Function Classification System (GMFCS); having spasticity at lower extremity 2 or less according to Modified Ashworth Scale, and being able to follow and accept verbal instructions. The exclusion criteria were having any orthopedic surgery or botulinum toxin injection in the past 6 months and having allergic reactions to the adhesive compound of KT.

Procedure

This study was designed as a randomized controlled trial. Twenty children (10 girls, 10 boys) were included in the study. The children were divided into two randomized groups using a computer program. Of the 20 participants, 11 were randomized to the taping group and 9 to the control group.

Measurements In the taping group, measurements were made at the beginning of the study, 30 minutes after the first tape was applied, and at the end of the 4th week. In the control group, measurements were made at the beginning of the study and at the end of the 4th week. The BTS G-Walk Spatiotemporal Gait Analysis System was administered by the third author (S. Ö.). All other measurements were administered by the same physiotherapist (S. N. K.). Gross motor function was classified using the GMFCS.

Body Structures and Functions Body composition was evaluated by body mass index (BMI) calculated with the following formula: weight in kilograms divided by the square of the height in meters. Balance was evaluated with the Pediatric Berg Balance Scale (PBBS).

Activity functioning Functionality was assessed using the Timed Up and Go test (TUG) and the Functional Mobility Scale (FMS). The TUG measures various components such as walking speed, postural control, functional mobility, and balance . The walking ability of the participants was evaluated with the Functional Mobility Scale at 3 different distances (5 meters-indoor, 50 meters-school, 500 meters-community). Inter-observer reliability of the FMS, which can reveal changes that cannot be detected with the GMFCS, was also demonstrated. Gross motor function was assessed using dimensions D and E of the Gross Motor Function Measurement (GMFM), which consists of standing, walking, running, and jumping. The GMFM is a valid, reliable, and sensitive method, which demonstrates the change in motor functions in children with CP and other disabilities via videotape recordings.

Gait parameters were assessed using the BTS G-Walk Spatiotemporal Gait Analysis System. In this system, the analysis results of the sensor attached to the L5-S1 level of the patient was transferred to a computer via Bluetooth. This system allows gait analysis by comparing the left and right extremities with normal values, and it also enables a 3-dimensional kinematic analysis of the pelvis. The track length was preset as 10 meters. The children with CP were asked to walk the 10-meter track three times. Three measurements were averaged in the analysis.

Participation Participation was assessed using the Canadian Occupational Performance Measure (COPM). The COPM is a client-centered outcome measure to identify and prioritize everyday issues that restrict individuals' participation in everyday life.

Intervention

Every group received routine traditional physiotherapy twice a week over the period of 4 weeks. This routine traditional treatment consisted of stretching, weight bearing, functional reaching, walking, and electrotherapy. Sessions were 40 minutes. The children in the taping group were taped 6 days per week for 4 weeks. The children were checked for allergies before applying the tape. A 5-cm tape was applied and kept in position for 3 days, and the region was then left to rest for 24 hours.

KT was applied to the gluteus maximus and gluteus medius muscles. The KT muscle facilitation technique was used to support and facilitate the function of the muscles. For the gluteus maximus, a "Y" tape was used. The child was placed in a side lying position and the beginning of the tape was applied to the origin of the muscle (center of the sacrum). The leg flexed and adducted, and the first tail was applied to enclose the lower part of the gluteus maximus muscle. The second tail was applied diagonally from the sacrum to the greater trochanter. For the gluteus medius muscle, 2 "I" tapes were applied. The first tape was applied from the spina iliaca anterior superior to the greater trochanter, the second tape was applied from the spina iliaca posterior superior to the greater trochanter. During the applications, the hip was adducted and extended, and all tape ends were applied without tension.

Statistical analysis Post-hoc power analysis was performed when 20 participants (11 in the taping group, 9 in the control group) were enrolled in our study. Power analysis was conducted using G*Power (version 3.0.10 Universitat Düsseldorf, Düsseldorf, Germany) to compare pairs of independent sample means. In the post-hoc power analysis, when the statistical significance of alpha was 5% and the confidence interval was 95%, the power of the study (1-β) was found to be 99%. The study was completed by deciding that a sufficient sample size was reached. The Statistical Package for the Social Sciences (SPSS) version 26 was used to analyze the obtained data. The level of significance was set at p<0.05. One-sample Kolmogorov-Smirnov Tests were used to evaluate distribution of variables before test selection. Descriptive analyses are presented using medians and the interquartile ranges for the non-normally distributed and ordinal variables. In the comparison of two independent nominal variables, while the Chi-Square Test was used, the Fisher Test was preferred according to the expected values in the table cells. The Mann-Whitney U test was used to compare non-normally distributed ordinal data in independent groups. The Wilcoxon Signed Ranks Test or the Friedman was used in dependent groups. The Student's t-test was used to compare normally distributed numerical data. Repeated Measures Anova was used to compare normally distributed numerical data in more than two dependent groups. Groups were compared with each other using the paired T test.

ELIGIBILITY:
Inclusion Criteria:

* having unilateral spastic CP
* being in an age between 6 years and 12 years;
* being classified in levels I or II of the Gross Motor Function Classification System (GMFCS); -having spasticity at lower extremity 2 or less according to Modified Ashworth Scale
* being able to follow and accept verbal instructions.

Exclusion Criteria:

* having any orthopedic surgery or botulinum toxin injection in the past 6 months
* having allergic reactions to the adhesive compound of Kinesio Taping

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Pediatric Berg Balance Scale (PBBS) | baseline and after 4 weeks
  Balance was evaluated with the Pediatric Berg Balance Scale (PBBS).On this scale minimum score is 0 and maximum score is 56. As the score increases, the balance improves. Between baseline and fourth week the balance change was assessed.
Timed Up and Go test (TUG) | baseline, 30 minutes after the first tape was applied, and at the end of the 4th week
  The TUG measures various components such as walking speed, postural control, functional mobility, and balance. Change in functionality was assessed between baseline, 30 minutes after the first taping, and at the fourth week.
Functional Mobility Scale (FMS) | baseline and after 4 weeks
  The walking ability of the participants was evaluated with the Functional Mobility Scale at 3 different distances (5 meters-indoor, 50 meters-school, 500 meters-community). Inter-observer reliability of the FMS, which can reveal changes that cannot be detected with the GMFCS, was also demonstrated.On this scale the minimum score is 1, and the maximum score is six. The higher the score, the better the functional status.Change in functionality was assessed between baseline and at the fourth week.
Gross Motor Function Measurement (GMFM) | baseline and after 4 weeks
  Gross motor function was assessed using dimensions D and E of the Gross Motor Function Measurement (GMFM), which consists of standing, walking, running, and jumping. The GMFM is a valid, reliable, and sensitive method, which demonstrates the change in motor functions in children with CP and other disabilities via videotape recordings. Minimum score is 0 and maximum score is 74. The higher the score, the better the functional status. Between baseline and fourth week the motor performance change was assessed.
BTS G-Walk Spatiotemporal Gait Analysis System | baseline, 30 minutes after the first tape was applied, and at the end of the 4th week
  Gait parameters were assessed using the BTS G-Walk Spatiotemporal Gait Analysis System. In this system, the analysis results of the sensor attached to the L5-S1 level of the patient was transferred to a computer via Bluetooth. This system allows gait analysis by comparing the left and right extremities with normal values, and it also enables a 3-dimensional kinematic analysis of the pelvis (11). The track length was preset as 10 meters. The children with CP were asked to walk the 10-meter track three times. Three measurements were averaged in the analysis. Change in gait parameters was assessed between baseline, 30 minutes after first taping and at the fourth week.
Canadian Occupational Performance Measure (COPM) | baseline and after 4 weeks
  Participation was assessed using the Canadian Occupational Performance Measure (COPM). The COPM is a client-centered outcome measure to identify and prioritize everyday issues that restrict individuals' participation in everyday life.There is no minimum maximum score on this scale. The pre- and post-treatment scores of the person are compared. Between baseline and fourth week the participation change was assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Seda Nur KEMER,PT, MSc, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No